CLINICAL TRIAL: NCT03872401
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Impact of Evolocumab on Major Cardiovascular Events in Patients at High Cardiovascular Risk Without Prior Myocardial Infarction or Stroke
Brief Title: Effect of Evolocumab in Patients at High Cardiovascular Risk Without Prior Myocardial Infarction or Stroke
Acronym: VESALIUS-CV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20170625; 2023-503673-38-00 (EU CTIS Number); 2018-004565-14 (EudraCT Number)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: High Cardiovascular Risk; No prior Myocardial Infarction stroke; >= 50 years of age (men); >= 55 years of age (women); lipid-lowering therapy
MeSH Terms: conditions — Coronary Disease; Multiple Endocrine Neoplasia Type 1 | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo subcutaneous injection once every 2 weeks (Q2W).
  Interventions: Drug: Placebo
- Evolocumab 140 mg Q2W (Experimental): Participants will receive 140 mg evolocumab by subcutaneous injection Q2W.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Administered subcutaneously using an autoinjector pen.
  Other Names: AMG 145; Repatha
  Arms: Evolocumab 140 mg Q2W
Drug: Placebo — Administered subcutaneously using an autoinjector pen.
  Arms: Placebo

SUMMARY:
This study will assess the effect of lowering low-density lipoprotein cholesterol (LDL-C) with evolocumab on major cardiovascular events in adults without a prior myocardial infarction (MI) or stroke who are at high risk of a cardiovascular event.

ELIGIBILITY:
Inclusion criteria:

* Age: Adult participants ≥ 50 (men) or ≥ 55 (women) to ˂ 80 years of age (either sex) and meeting lipid criteria.
* Lipid Criteria: Low-density lipoprotein cholesterol (LDL-C) ≥ 90 mg/dL (≥ 2.3 mmol/L) or non high-density lipoprotein cholesterol (non-HDL)-C ≥ 120 mg/dL (≥ 3.1 mmol/L), or apolipoprotein B ≥ 80 mg/dL (≥ 1.56 µmol/L).

  3.Diagnostic evidence of at least one of the following (A-D) at screening:

A.Significant coronary artery disease (CAD) meeting at least 1 of the following criteria:

* History of coronary revascularization with multi-vessel coronary disease as evidenced by any of the following:

  1. percutaneous coronary intervention (PCI) of 2 or more vessels, including branch arteries,
  2. PCI or coronary artery bypass grafting (CABG) with residual 50% stenosis in a separate, unrevascularized vessel, or
  3. multi-vessel CABG 5 years or more prior to screening.
* Significant coronary disease without prior revascularization as evidenced by either a ≥70% stenosis of at least 1 coronary artery, ≥50% stenosis of 2 or more coronary arteries, or ≥50% stenosis of the left main coronary artery.
* known coronary artery calcium score ≥100 in participants without a coronary artery revascularization prior to randomization.

B. Significant atherosclerotic cerebrovascular disease meeting at least 1 of the following criteria:

* prior transient ischemic attack with ≥50% carotid stenosis.
* internal or external carotid artery stenosis of ≥70% or 2 or more ≥50% stenoses.
* prior internal or external carotid artery revascularization.

C. Significant peripheral arterial disease meeting at least 1 of the following criteria:

* ≥50% stenosis in a limb artery.
* history of abdominal aorta treatment (percutaneous and surgical) due to atherosclerotic disease.
* ankle brachial index (ABI) <0.85.

D. Diabetes mellitus with at least 1 of the following:

* known microvascular disease, defined by diabetic nephropathy or treated retinopathy. Diabetic nephropathy defined as persistent microalbuminuria (urinary albumin to creatinine ratio ≥30mg/g) and/or persistent estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m^2 that is not reversible due to an acute illness.
* chronic daily treatment with an intermediate or long-acting insulin.
* diabetes diagnosis ≥10 years ago.

  •At least 1 of the following 1 high-risk criteria (most recent lab values within 6 months prior to screening, as applicable):
* Polyvascular disease, defined as coronary, carotid, or peripheral artery stenosis ≥50% in a second distinct vascular location in a participant with coronary, cerebral or peripheral arterial disease (A, B, or C above).
* Presence of either diabetes mellitus or metabolic syndrome in a participant with coronary, cerebral, or peripheral artery disease (A, B, or C above).
* At least 1 coronary, carotid, or peripheral artery residual stenosis of ≥50% in a participant with diabetes meeting inclusion criterion (D above).
* LDL-C ≥130 mg/dL (≥3.36 mmol/L), OR non-HDL-C ≥160 mg/dL (≥4.14 mmol/L), OR apolipoprotein B ≥120 mg/dL (2.3 µmol/L) if available.
* Lipoprotein (a) >125 nmol/L (50 mg/dL).
* Known familial hypercholesterolemia.
* Family history of premature coronary artery disease defined as an MI or CABG in the participant's father or brother at age <55 years or an MI or CABG in the participant's mother or sister at age <60 years.
* High sensitive c-reactive protein (hsCRP) ≥3.0 mg/L in the absence of an acute illness.
* Current tobacco use.

  -≥65 years of age.
* Menopause before 40 years of age.
* eGFR 15 to <45 mL/min/1.73 m^2.
* Coronary artery calcification score ≥300 in a participant without a coronary revascularization prior to randomization.

Exclusion criteria

* MI or stroke prior to randomization.
* CABG ˂ 3 months prior to screening.
* eGFR ˂ 15 mL/min/1.73 m^2.
* Uncontrolled or recurrent ventricular tachycardia in the absence of an implantable-cardioverter defibrillator.
* Atrial fibrillation or atrial flutter not on anticoagulation therapy (vitamin K antagonist, heparin, low molecular weight heparin, fondaparinux,or non-Vitamin K antagonist oral anticoagulant).
* Triglycerides ≥ 500 mg/dL (5.7 mmol/L) measured up to 3 months prior to screening. The most recent results must be used.
* Last measured left-ventricular ejection fraction ˂ 30% or New York Heart Association (NYHA) Functional Class III/IV.
* Planned arterial revascularization.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12301 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Time to Coronary Heart Disease Death, Myocardial Infarction, or Ischemic Stroke | From randomization; for approximately a median of 4.5 years
  Time to coronary heart disease (CHD) death, myocardial infarction (MI), or ischemic stroke, whichever occurs first.
Time to Coronary Heart Disease Death, Myocardial Infarction, Ischemic Stroke, or Any Ischemia-driven Arterial Stroke | From randomization; for approximately a median of 4.5 years
  Time to CHD death, MI, ischemic stroke, or any ischemia-driven arterial revascularization, whichever occurs first.

SECONDARY OUTCOMES:
Time to MI, Ischemic Stroke, or Any Ischemia-driven Arterial Revascularization | From randomization; for approximately a median of 4.5 years
Time to CHD Death, MI, or Any Ischemia-driven Arterial Revascularization | From randomization; for approximately a median of 4.5 years
Time to Cardiovascular Death, MI, or Ischemic Stroke | From randomization; for approximately a median of 4.5 years
Time to CHD Death or MI | From randomization; for approximately a median of 4.5 years
Time to Myocardial Infarction | From randomization; for approximately a median of 4.5 years
Time to Any Ischemia-driven Arterial Revascularization | From randomization; for approximately a median of 4.5 years
Time to CHD Death | From randomization; for approximately a median of 4.5 years
Time to Cardiovascular Death | From randomization; for approximately a median of 4.5 years
Time to All Cause of Death | From randomization; for approximately a median of 4.5 years
Time to Ischemic Stroke | From randomization; for approximately a median of 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (849):
- United States (145):
  - North Alabama Research Center LLC, Athens, Alabama
  - Cardiovascular Associates, Birmingham, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - Mobile Heart Specialists PC, Mobile, Alabama
  - Arkansas Cardiology, Little Rock, Arkansas
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Cardiovascular Research Foundation of Southern California, Beverly Hills, California
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - West Coast Research LLC, Dublin, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Covigilant Research, LLC, Riverside, California
  - Sierra Clinical Research, Roseville, California
  - Center for Clinical Trials of Sacramento Inc, Sacramento, California
  - Harbor University of California Los Angeles Medical Center, Torrance, California
  - Optumcare Colorado Springs LLC, Colorado Springs, Colorado
  - University of Colorado Memorial Health System, Colorado Springs, Colorado
  - New West Physicians, Golden, Colorado
  - South Denver Cardiology Associates, Littleton, Colorado
  - Cardiology Associates of Fairfield County, PC, Stamford, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Bay Area Cardiology, Brandon, Florida
  - Nature Coast Clinical Research LLC, Crystal River, Florida
  - Daytona Heart Group, Daytona Beach, Florida
  - Cardiology Research Associates, Daytona Beach, Florida
  - Complete Health Research, DeLand, Florida
  - Cohen Medical Associates PA, Delray Beach, Florida
  - Jellinger and Lerman MD PA dba The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - George E Platt MD, Green Cove Springs, Florida
  - Research Physicians Network Alliance, Hollywood, Florida
  - University of Florida and Shands Hospital, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - First Coast Cardiovascular Institute PA, Jacksonville, Florida
  - Baptist Health Research Institute, Jacksonville Beach, Florida
  - Gad Research Center, Miami, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Ocala Research Institute, Inc, Ocala, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Florida Cardiology Group, Winter Park, Florida
  - The Florida Lipid Institute, Winter Park, Florida
  - NSC Research, Johns Creek, Georgia
  - Kootenai Heart Clinics, LLC, Coeur d'Alene, Idaho
  - Northwest Heart Clinical Research LLC, Arlington Heights, Illinois
  - Deaconess Clinic, Evansville, Indiana
  - LaPorte County Institute for Clinical Research, Michigan City, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - The University of Iowa College of Public Health, Iowa City, Iowa
  - MercyOne Iowa Heart Center, West Des Moines, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Saint Elizabeth Covington, Covington, Kentucky
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Grace Research LLC, Bossier City, Louisiana
  - Horizon Research Group of Opelousas LLC, Eunice, Louisiana
  - Louisiana Heart Center, Hammond, Louisiana
  - Barnum Medical Research, Natchitoches, Louisiana
  - Grace Research LLC, Shreveport, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Southern Maine Health Care, Biddeford, Maine
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants LLC, Beltsville, Maryland
  - TidalHealth Peninsula Regional, Inc, Salisbury, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Charles River Medical Associates, Framingham, Massachusetts
  - East Mountain Medical Associates, PC, Great Barrington, Massachusetts
  - Baystate Health Center, Springfield, Massachusetts
  - Ahmed Arif Medical Research Center LLC, Flint, Michigan
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - Rajendra H Mehta, MD, PC, Jackson, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint Marys Medical Center, Duluth, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - HealthEast Medical Research Institute, Saint Paul, Minnesota
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Mercy Research, St Louis, Missouri
  - Great Falls Clinic LLP, Great Falls, Montana
  - Bryan Heart, Lincoln, Nebraska
  - Nebraska Western Iowa Health Care System, Omaha, Nebraska
  - Palm Research Center Inc, Las Vegas, Nevada
  - Virtua Health, Inc., Voorhees Township, New Jersey
  - Healthwise Medical Associates, Brooklyn, New York
  - Trinity Medical Western New York, PC, Cheektowaga, New York
  - WMCHealth Heart and Vascular Institute Kingston Division of Cardiology, Kingston, New York
  - Northwell Health Physician Partners Cardiology, Manhasset, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Northwell Health Lenox Hill Heart and Vascular, New York, New York
  - Hudson Valley Cardiovascular Physicians PC, Poughkeepsie, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Division of Cardiovascular Research at Peconic Bay Medical Center, Southampton, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Moses H Cone Memorial Hospital, Greensboro, North Carolina
  - Crossroads Clinical Research Inc, Mooresville, North Carolina
  - Piedmont Medical Group Research of Rocky Mount, Rocky Mount, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - North Ohio Heart Center, Elyria, Ohio
  - Sanjay Vora Research LLC, Marion, Ohio
  - North Ohio Heart Center-Sandusky, Sandusky, Ohio
  - Heart House Research Foundation, Springfield, Ohio
  - Intend Research, Norman, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Capital Area Research LLC, Camp Hill, Pennsylvania
  - Geisinger Holy Spirit, Camp Hill, Pennsylvania
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - Lycoming Internal Medicine Inc, Jersey Shore, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Cardiology Consultants of Philadelphia CCP, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Pharmacorp Clinical Trials Inc, Charleston, South Carolina
  - Piedmont Research Partners, Fort Mill, South Carolina
  - Tribe Clinical Research LLC DBA Mountain View Clinical Research, Greenville, South Carolina
  - Main Street Physicians Care Waterway, Little River, South Carolina
  - The Diabetes Center, Murrells Inlet, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Parkway Cardiology Associates, Oak Ridge, Tennessee
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Humble Cardiology Associates, Kingwood, Texas
  - Texas Cardiology Associates of Houston, Kingwood, Texas
  - Texas Institute for Kidney and Endocrine Disorders, Lufkin, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Southern Endocrinology Associates PA, Mesquite, Texas
  - Permian Research Foundation, Odessa, Texas
  - South Texas Cardiovascular Consultants PLLC, San Antonio, Texas
  - Mercury Medical Conversions LTD, San Antonio, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Alpine Research Organization, Farmington, Utah
  - Suffolk Multispecialty Research LLC, Suffolk, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Multicare Institute for Research and Innovation, Puyallup, Washington
  - Universal Research Group LLC, Tacoma, Washington
  - Aspirus Research Institute, Wausau, Wisconsin
- Argentina (33):
  - Instituto de Investigaciones Clinicas Bahia Blanca, Bahía Blanca, Buenos Aires
  - Stat Research, CABA, Buenos Aires
  - Cinme - Centro de Investigaciones Metabolicas, CABA, Buenos Aires
  - Ciprec - Centro de Investigacion y Prevencion Cardiovascular, CABA, Buenos Aires
  - Consultorio Medico Dr Litvak Bruno, CABA, Buenos Aires
  - Centro de Especialidades Medicas - Cemedic, CABA, Buenos Aires
  - Centro Medico Laura Maffei, CABA, Buenos Aires
  - Cardiología Palermo, CABA, Buenos Aires
  - Cedic - Centro de Investigacion Clinica, CABA, Buenos Aires
  - Centro Medico Dra De Salvo, CABA, Buenos Aires
  - Fundacion Respirar, CABA, Buenos Aires
  - Instituto de Investigaciones Metabolicas - Idim, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Universitario Fundacion Favaloro, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Icba - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Glenny Corp SA, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - Ciad - Consultorio Integral de Atencion al Diabetico, Morón, Buenos Aires
  - Dim Clinica Privada, Ramos Mejía, Buenos Aires
  - Instituto de Investigaciones Clinicas de San Nicolas, San Nicolás de los Arroyos, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Clinica Privada del Prado, Córdoba, Córdoba Province
  - Clinica Fusavim Privada SRL, Villa María, Córdoba Province
  - Sanatorio Santa Rosa Srl, Santa Rosa, La Pampa Province
  - Instituto de Investigaciones Clínicas Rosario-Sanatorio Delta, Rosario, Santa Fe Province
  - Sanatorio Plaza, Rosario, Santa Fe Province
  - Centro Modelo de Cardiologia, San Miguel de Tucumán, Tucumán Province
  - Clinical Mayo de Urgencias Medicas Cruz Blanca SRL, San Miguel de Tucumán, Tucumán Province
  - Instituto de Cardiologia de Corrientes Juana Francisca Cabral, Corrientes
  - Instituto Medico DAMIC - Fundacion Rusculleda, Córdoba
  - Cordis Sa, Salta
  - Clinica El Castano, San Juan
  - Instituto Cardiovascular San Luis, San Luis
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- Australia (22):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Heartcare Partners, Auchenflower, Queensland
  - Bundaberg Cardiology, Bundaberg, Queensland
  - Holdsworth House Medical Brisbane, Fortitude Valley, Queensland
  - Core Research Group Pty Ltd, Milton, Queensland
  - Heart and Vascular Research, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - SA Heart, Ashford, South Australia
  - Adelaide Cardiology Practice - Leabrook Clinic, Leabrook, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - HeartCare Victoria - Berwick, Berwick, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - The Cardiologists Proprietary Limited, Epping, Victoria
  - Barwon Health Geelong Hospital, Geelong, Victoria
  - GenesisCare Ringwood, Ringwood, Victoria
  - Curtin University Centre of Clinical Research and Education, Bentley, Western Australia
  - HeartCare Western Australia - Joondalup, Joondalup, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Dr Heart Pty Ltd, Woolloongabba
- Austria (10):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Klinik Landstrasse, Vienna
  - Zentrum fuer klinische Studien - Dr Hanusch GmbH, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
  - Klinik Ottakring, Vienna
- Belgium (15):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - Onze Lieve Vrouw Ziekenhuis - campus Aalst, Aalst
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - AZ Sint Blasius, Dendermonde
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - Medif sprl, Gozée
  - Dokter Mortelmans bvba, Ham
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Medilink sprl, Linkebeek
  - Centre Hospitalier Universitair Ambroise Pare, Mons
  - Maria Ziekenhuis Noord-Limburg, Overpelt
  - Testumed vzw, Tessenderlo
- Brazil (20):
  - Centro de Pesquisas em Diabetes e Doencas Endocrino Metabolicas, Fortaleza, Ceará
  - Centro de Pesquisa Clinica do Brasil, Brasília, Federal District
  - Cardresearch Cardiologia Assistencial de Pesquisa, Belo Horizonte, Minas Gerais
  - Fundaçao Hospitalar Sao Francisco de Assis, Belo Horizonte, Minas Gerais
  - Eurolatino Pesquisas Medicas, Uberlândia, Minas Gerais
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul, Paraná
  - Quanta Diagnosticos e Terapia, Curitiba, Paraná
  - Puc Trials - Núcleo de Pesquisa Clínica da Escola de Medicina da Pucpr/Epicenter, Curitiba, Paraná
  - Nucleo de Pesquisa Clinica, Curitiba, Paraná
  - Núcleo de Pesquisa em Cirurgia Vascular, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - AngioCor Blumenau, Blumenau, Santa Catarina
  - Centro Especializado em Cardiologia, Campinas, São Paulo
  - Instituto de Pesquisa Clinica de Campinas, Campinas, São Paulo
  - Instituto do Coracao de Marilia, Marília, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Centro de Pesquisas Clinicas Cpclin, São Paulo, São Paulo
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
  - Instituto do Coracao do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Bulgaria (19):
  - Ambulatory for special outpatient medical aid in Cardiology-Private Practice Dr Elena Dotcheva EOOD, Burgas
  - Multiprofile Hospital for Active Treatment - Haskovo AD, Haskovo
  - Specialty Hospital for Active treatment in Cardiology Sveti Georgi - Pernik OOD, Pernik
  - Medical Center Medconsult OOD, Pleven
  - University Multiprofile Hospital for Active Treatment Dr Georgi Stranski EAD, Pleven
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Multiprofile Hospital for Active Treatment- Medical Complex- Sveti Ivan Rilski EOOD, Plovdiv
  - Fifth Multiprofile Hospital for Active Treatment - Sofia EAD, Sofia
  - National Multiprofile Transport Hospital Tzar Boris III, Sofia
  - Medical Center for Specialized Medical Care of Cardiovascular Diseases OOD, Sofia
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
  - Medical Center Excelsior OOD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N I Pirogov EAD, Sofia
  - Diagnostic-Consultative Center Convex EOOD, Sofia
  - Medical Center Kalimat EOOD, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Anna Sofia AD, Sofia
  - Medical Center Orpheus OOD, Stara Zagora
  - Multiprofile Regional Hospital for Active Treatment Dr Stefan Cherkezov AD, Veliko Tarnovo
- Canada (36):
  - LMC Clinical Research Incorporated, Calgary, Alberta
  - SMH Cardiology Clinical Trials Incorporated, Surrey, British Columbia
  - Dr T G Elliott Incorporated - BC Diabetes, Vancouver, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - G A Research Associates Limited, Moncton, New Brunswick
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre, Halifax Infirmary, Halifax, Nova Scotia
  - Heart Health Institute, Ajax, Ontario
  - LMC Clinical Research Incorporated, Barrie, Ontario
  - LMC Clinical Research Incorporated, Brampton, Ontario
  - Brampton Clinical Trials, Brampton, Ontario
  - LMC Clinical Research Incorporated Thornhill, Concord, Ontario
  - LMC Clinical Research Incorporated, Etobicoke, Ontario
  - Hamilton Health Sciences Hamilton General Hospital, Hamilton, Ontario
  - Western Centre for Public Health and Family Medicine - Western University, London, Ontario
  - My Endo Diabetes and Endocrinology Center, Markham, Ontario
  - LMC Clinical Research Incorporated, Nepean, Ontario
  - Partners in Advanced Cardiac Evaluation, Newmarket, Ontario
  - SKDS Research Incorporated, Newmarket, Ontario
  - Oakville Cardiovascular Research, Oakville, Ontario
  - Dr James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Bluewater Clinical Research Group Incorporated, Sarnia, Ontario
  - Heart Health Institute Research Incorporated, Scarborough Village, Ontario
  - Corcare Cardiovascular Research, Scarborough Village, Ontario
  - Womens College Hospital, Toronto, Ontario
  - North York Diagnostic and Cardiac Centre, Toronto, Ontario
  - Office of Dr Louis Yao, Weston, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Manna Research Incorporated, Lévis, Quebec
  - Clinique Sante Cardio MC, Montreal, Quebec
  - Institut de recherches cliniques de Montreal, Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital, Montreal, Quebec
  - Applied Medical Informatics Research Incorporated, Montreal, Quebec
  - Clinique des Maladies Lipidiques de Quebec Incorporated, Québec, Quebec
  - Centre intégré de santé et de services sociaux (CISSS) des Laurentides - Unité de recherche clini, Saint-Jérôme, Quebec
- Czechia (54):
  - MUDr Igor Karen, Benátky nad Jizerou
  - Jessenia as, Nemocnice Beroun, Beroun
  - Medicentrum Beroun sro, Beroun
  - Medicus Services sro, Brandýs nad Labem
  - Amkardia sro, Brno
  - CCR Brno sro, Brno
  - Centrum pro zdravi sro, Brno
  - Kardiologicka ambulance Brno sro, Brno
  - Fakultni nemocnice Brno, Brno
  - Vojenska nemocnice Brno, Brno
  - prof MUDr Lubomir Elbl, CSc, Kardiologicka ambulance, Brno
  - Edumed sro, Kardiologicka ambulance, Broumov
  - Cevni centrum Ceske Budejovice sro, České Budějovice
  - Dika centrum sro, Havirov - Mesto
  - Clinical Trial Center Hodonin sro, Hodonín
  - Kardio Holesov sro, Holešov
  - MUDr Ladislava Harrerova, kardiologicka ordinace, Hradec Králové
  - Karlovarska krajska nemocnice, Karlovy Vary
  - Oblastni nemocnice Kladno as, Kladno
  - Kardio Michal Cepelak sro, Klatovy IV
  - Oblastni nemocnice Kolin as, Kolin III
  - Krajska nemocnice Liberec as, Liberec
  - KardioBusak sro, Louny
  - Kardio Pudich s.r.o., Ludgeřovice
  - Vseobecna intermi ambulance sro, Milevsko
  - MUDr Zbynek Kosek, kardiologicka ambulance sro, Mladá Boleslav
  - Pozdisek sro, Kardiologicka ambulance, Mohelnice
  - CCR Ostrava sro, Ostrava
  - Mestska nemocnice Ostrava, Ostrava
  - Benedor sro - Kardiologicka, cevni a interni ambulance, Ostrava - Poruba
  - Kardiologicka a angiologicka ambulance, Ostrava-Dubina
  - Center for Clinical Research Pardubice, sro, Pardubice
  - Nemocnice Pardubickeho kraje as, Pardubice
  - Kardiologie v sadech sro, Pilsen
  - Ordinace pro choroby srdce a cev, Prague
  - Diabet2 sro, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - CCR Prague sro, Prague
  - Thomayerova nemocnice, Prague
  - Milan Kvapil sro, Prague
  - Fakultni nemocnice v Motole, Prague
  - Interni a kardiologicka ordinace, Prague
  - Endokrinologie Cerny Most sro, Prague
  - Kardiologie Cor sro, Praha 10 - Zabehlice
  - Kardiologicke centrum MUDr Janky Skrobakove sro, Praha 5 - Smichov
  - Kardio Vaclavik sro, Interni a kardiologicka ambulance, Přerov
  - Vestra Clinics sro, Rychnov nad Kněžnou
  - Nemocnice Pardubickeho kraje as, Svitavska nemocnice, Svitavy
  - AeskuLab ks, Lipidova poradna, Teplice
  - Nemocnice Podlesi as, Třinec
  - Clinical Trials Service sro, Uherské Hradiště
  - Interni ambulance, Uherské Hradiště
  - Lekarsky dum Ormiga, Zlín
  - KIGE sro, Znojmo
- Denmark (16):
  - Aalborg Hospital, Aalborg
  - Center for Clinical and Basic Research Aalborg, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Centre for Clinical and Basic Research Ballerup, Ballerup Municipality
  - Sydvestjysk Sygehus, Esbjerg
  - Sanos Clinic, Herlev
  - Steno Diabetes Center, Herlev
  - Regionhospitalet Herning, Herning
  - Hillerod Hospital, Hillerød
  - Kolding Sygehus, Kolding
  - Amager Hospital, København S
  - Rigshospitalet Kobenhavn, København Ø
  - Regionshospitalet Silkeborg, Silkeborg
  - Svendborg Sygehus, Svendborg
  - Center for Clinical and Basic Research Vejle, Vejle
  - Regionshospitalet Viborg, Viborg
- Estonia (4):
  - Liina Viitas OU, Pärnu
  - Center for Clinical and Basic Research Tallinn, Tallinn
  - Dr Arvo Rosenthal LLC, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
- Finland (10):
  - Helsinki University Central Hospital, Helsinki
  - GERI-MED Oy, Helsinki
  - Pohjois-Karjalan keskussairaala, Joensuu
  - Terveystalo Jyvaskyla, Jyväskylä
  - Studycor Oy, Jyväskylä
  - Satucon Oy/Kuopion tyoterveys, Kuopio
  - University of Eastern Finland, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Terveystalo Pulssi, Turku
- France (27):
  - Centre Hospitalier Universitaire Amiens - Hopital Sud, Amiens
  - Hospices Civils de Lyon Groupement Hospitalier Est, Hopital Louis Pradel, Bron
  - Centre Hospitalier Universitaire de Caen - Hôpital Côte de Nacre, Caen
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Universitaire de Dijon - Hopital Francois Mitterrand, Dijon
  - Groupement Hospitalier Mutualiste, Grenoble
  - Centre Hospitalier Universitaire de Grenoble - Hopital Nord Michallon, Grenoble
  - Centre Hospitalier de Versailles - Hopital Andre Mignot, Le Chesnay
  - Hopital Louis Pasteur, Le Coudray
  - Centre Hospitalier Régional Universitaire de Lille - Institut Coeur Poumon, Lille
  - Centre Hospitalier Universitaire de Lyon - Hopital Edouard Herriot, Lyon Cédex 3
  - Hopital Saint-Joseph, Marseille
  - Centre Hospitalier Universitaire de Marseille - Hôpital de la Timone, Marseille
  - Centre Hospitalier Regional Universitaire de Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Universitaire de Nantes - Hopital Guillaume et Rene Laennec, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Centre Hospitalier Universitaire de Nimes, Nîmes
  - Hopital Saint Antoine, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Centre Hospitalier de Pau - Hopital Francois Mitterrand, Pau
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Clinique Saint Hilaire, Rouen
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
  - Polyclinique Vauban, Valenciennes
- Germany (31):
  - Universitaets-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik Forschungs GmbH, Bad Neuheim
  - Klinische Forschung Berlin GbR, Berlin
  - Charite Universitätsmedizin Berlin, Charité Campus Virchow-Klinikum, Berlin
  - Kardiologisch - Angiologische Praxis - Herzzentrum Bremen, Bremen
  - Sankt-Johannes-Hospital, Dortmund
  - Cardiologicum Dresden und Pirna, Dresden
  - Diabetologische Gemeinschaftspraxis Dr Schaper und Dr Faulmann, Dresden
  - Universitaetsklinikum Carl Gustav Carus, Medizinische Klinik und Poliklinik III, Dresden
  - Klinikum und Fachbereich Medizin Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main
  - Clin Phenomics GmbH Co KG, Frankfurt am Main
  - Medizinisches Versorgungszentrum im Altstadt-Carree Fulda, Fulda
  - Cardiologicum Hamburg, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Ambulantes Herzzentrum Kassel, Kassel
  - Universitätsklinikum Leipzig, Leipzig
  - Otto von Guericke Universität Magdeburg, Magdeburg
  - Johannes Gutenberg Universitaet Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Praxis Doktor Jens Taggeselle, Markleeberg
  - Deutsches Herzzentrum München des Freistaates Bayern, München
  - Herz Gefaess Zentrum Nymphenburg, München
  - Universitaetsklinikum Muenster, Münster
  - Kardiologische Gemeinschaftspraxis Papenburg, Papenburg
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - Universitätsklinikum Regensburg, Regensburg
  - CardioConsil GmbH, Rostock
  - I Medizinische Klinik Gesundheitsverbund Landkreis Konstanz, Singen
  - Universitätsklinikum Ulm, Ulm
  - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen
  - Forschungszentrum Ruhr, Witten
- Greece (15):
  - General Hospital of Athens Evaggelismos, Athens
  - Athens Naval Hospital, Athens
  - General Hospital of Athens Georgios Gennimatas, Athens
  - General Hospital of Athens Ippokrateio, Athens
  - General Hospital of Athens Laiko, Athens
  - Alexandra Hospital, Athens
  - Konstantopoulio - Agia Olga Hospital of Nea Ionia, Athens
  - Hygeia Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - University Hospital of Larissa, Larissa
  - Ahepa University Hospital, Thessaloniki
  - General Hospital of Thessaloniki Ahepa, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
  - Interbalkan Medical Center, Thessaloniki
- Hungary (37):
  - Lausmed Kft, Baja
  - Allami Szivkorhaz Balatonfured, Balatonfüred
  - Balatonmariafurdo Kozseg Onkormanyzatanak Haziorvosi Rendeloje, Balatonkeresztúr
  - Med-Edu Bt, Ballószög
  - Grof Tisza Istvan Korhaz, Berettyóújfalu
  - Dr Lakatos Ferenc Private Cardiology Practice, Békéscsaba
  - Betegapolo Irgalmas Rend - Budai Irgalmasrendi Korhaz, Budapest
  - Clinexpert Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Semmelweis Egyetem Varosmajori Sziv- es Ergyogyaszati Klinika, Budapest
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Budapest
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Semmelweis Egyetem, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Zugloi Egeszsegugyi Szolgalat, Budapest
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - Erzsebet Gondozohaz, Gödöllő
  - Bugat Pal Korhaz, Gyöngyös
  - Pharma4 Trial Kft, Gyöngyös
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - BKS Research Kft, Hatvan
  - Bacs-Kiskun Megyei Korhaz Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar Oktato Korhaza, Kalocsa
  - Selye Janos Korhaz, Komárom
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - CRU Hungary Kft, Miskolc
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Soproni Erzsebet Oktato Korhaz es Rehabilitacios Intezet, Sopron
  - Szegedi Tudomanyegyetem Szent Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Csongrad Megyei Dr Bugyi Istvan Korhaz, Szentes
  - Praxispont Belvarosi Maganegeszsegugyi Kozpont, Székesfehérvár
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Belvarosi Egeszseghaz Kft, Zalaegerszeg
- Iceland (2):
  - Hjartamidstodin, Kopavogur
  - Landspitali, Reykjavik
- Italy (16):
  - Ospedale Muscatello, Augusta
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero Universitaria di Bologna Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - Universita degli Studi Gabriele D Annunzio di Chieti e Pescara, Chieti
  - Fondazione Toscana Gabriele Monasterio Ospedale del Cuore G Pasquinucci, Massa
  - IRCCS Ospedale San Raffaele, Milan
  - Centro Cardiologico Monzino, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Presidio Ospedaliero Santa Maria delle Grazie, Pozzuoli
  - Policlinico Universitario Campus Biomedico, Roma
  - Azienda Ospedaliera Sant Andrea, Roma
  - IRCCS Policlinico San Donato, San Donato Milanese
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliero Universitaria Integrata di Udine, Udine
- Latvia (5):
  - Daugavpils Regional Hospital, Daugavpils
  - Dace Teterovska Doctor Practice in Endocrinology, Ogre
  - Inga Jasinkevica Cardiologist Practice, Ogre
  - Pauls Stradins Clinical University Hospital, Riga
  - Outpatient Clinic Veselibas Centrs 4, Riga
- Lithuania (7):
  - Klinikiniai sprendimai, UAB, Alytus
  - Klinikiniai sprendimai, UAB, Kaunas
  - Saules Seimos Medicinos Centras, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics Public Institution, Kaunas
  - Kardiologijos ir reabilitacijos klinika, UAB, Klaipėda
  - Siauliai Republican Hospital, Public Institution, Šiauliai
  - Vilnius University Hospital Santaros Clinic Public Institution, Vilnius
- Mexico (6):
  - Clinstile SA de CV, Cd de Mexico, Mexico City
  - Unidad Biomedica Avanzada Monterrey, Monterrey, Nuevo León
  - Centro de Estudios Clinicos de Queretaro, Querétaro City, Querétaro
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada SC, Culiacán, Sinaloa
  - Centro de investigacion Cardiometabolica, Aguascalientes
  - Scientia Investigacion Clinica Sc, Chihuahua City
- Netherlands (52):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Emotional Brain, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Van Weel Bethesda Ziekenhuis, Dirksland
  - Albert Schweitzer Ziekenhuis location Dordwijk, Dordrecht
  - Albert Schweitzer Ziekenhuis, Locatie Dordwijk, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Treant Zorggroep, locatie Scheper ziekenhuis Emmen, Emmen
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Sint Jansdal Ziekenhuis, Harderwijk
  - Zuyderland Medisch Centrum, Heerlen
  - Elkerliek Ziekenhuis, Helmond
  - Tergooi, Hilversum
  - Bethesda Diabetes Research Center, Hoogeveen
  - Dijklander Ziekenhuis Hoorn, Hoorn
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Isala Diaconessenhuis, Meppel
  - Sint Antonius Ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Radboudumc, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Franciscus Gasthuis, Rotterdam
  - Praktijk Soerland, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Franciscus Vlietland, Schiedam
  - D&A Research and Genetics, Sneek
  - Haga Ziekenhuis, The Hague
  - Huisartsenpraktijk Rambharose, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Elisabeth-Tweesteden Ziekenhuis, Tilburg
  - Ziekenhuis Bernhoven, Uden
  - Diakonessenhuis, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - Zaans Medisch Centrum, Zaandam
  - Albert Schweitzer Ziekenhuis, Zwijndrecht
  - Dokters van Nederhoven, Zwijndrecht
  - Isala Klinieken, Zwolle
- Poland (52):
  - Szpital Uniwersytecki nr 1 im dr Antoniego Jurasza w Bydgoszczy, Bydgoszcz
  - American Heart of Poland Sa Malopolskie Centrum Sercowo-Naczyniowe PAKS - Chrzanow, Chrzanów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Copernicus Podmiot Leczniczy Sp zoo, Gdansk
  - NZOZ Srodmiescie Spzoo, Gdynia
  - Marek Piepiorka Gabinet Kardiologiczno-Internistyczny, Gdynia
  - Spolka Cywilna Medicina, Giżycko
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni im swietego Jana Pawla II, Grodzisk Mazowiecki
  - Biokinetica SA, Józefów
  - Centrum Medyczne Pratia Katowice, Katowice
  - Specjalistyczna Poradnia Kardiologiczna i Nadcisnienia Tetniczego Beata Wozakowska-Kaplon, Kielce
  - Wojewodzki Szpital Zespolony w Kielcach, Kielce
  - Ewa Mirek-Bryniarska Specjalistyczna Praktyka Lekarska, Krakow
  - Zespol Przychodni Specjalistycznych Diab-End-Cor Sp z oo, Krakow
  - Krakowskie Centrum Medyczne Spzoo, Krakow
  - CARINTART Sp zoo Krakowskie Centrum Diagnostyczno-Kliniczne, Krakow
  - Intercard Spzoo Centrum Kardiologii Inwazyjnej Elektroterapii i Angiologii w Krosnie, Krosno
  - Wojewodzki Specjalistyczny Szpital im dr Wladyslawa Bieganskiego w Lodzi, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Miedziowe Centrum Zdrowia Spolka Akcyjna, Lubin
  - CenterMed Lublin Spzoo, Lublin
  - Clinical Best Solutions Sp zoo Spolka komandytowa Gabinet Lekarski, Lublin
  - Ko-med Centra Kliniczne Lublin II, Lublin
  - NZOZ Twoja Przychodnia Spzoo, Lublin
  - Szpital Swietej Anny w Miechowie, Miechów
  - Podhalanski Szpital Specjalistyczny im Jana Pawla II w Nowym Targu, Nowy Targ
  - Centrum Medyczne Pulawska spzoo Centrum Medyczne Pulawska NZOZ, Piaseczno
  - Clinical Research Center Spzoo Medic-R Spolka Komandytowa, Poznan
  - KO-MED Centra Kliniczne Spzoo KO-MED Centra Kliniczne Pulawy, Puławy
  - NZOZ Specjalistyczna Przychodnia Lekarska Medikard, Płock
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek Henryk Rudzki spolka jawna, Ruda Śląska
  - Clinical Best Solutions Spolka z ograniczona odpowiedzialnoscia Spolka komandytowa, Siedlce
  - ETG Network Spzoo, Skierniewice
  - KO-MED Centra Kliniczne Spzoo KO-MED Centra Kliniczne Staszow, Staszów
  - Indywidualna Specjalistyczna Praktyka Lekarska, Szczecin
  - Tomasz Blicharski Lubelskie Centrum Diagnostyczne, Świdnik
  - Centrum Szybkiej Diagnostyki Kardiologicznej Kardiomed M Zabowka E Zabowka Spolka cywilna, Tarnów
  - Medical Trials Institute Spzoo, Torun
  - Prywatne Centrum Kardiologii, Torun
  - Wojewodzki Szpital Zespolony im Ludwika Rydygiera w Toruniu, Torun
  - Centrum Medyczne Amed Warszawa Zoliborz, Warsaw
  - Centrum Medyczne Pratia Warszawa, Warsaw
  - Clinical Best Solutions Sp zoo Spolka komandytowa, Warsaw
  - Instytut Psychiatrii i Neurologii, Warsaw
  - Szpital Grochowski imienia Doktora medycyny Rafala Masztaka Spzoo, Warsaw
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej w Wegrowie, Węgrów
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Wroclaw
  - Centrum Kardiologiczne Pro Corde Spzoo Centrum Kardiologicne Pro Corde Wroclaw, Wroclaw
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw
  - Medicor Plus Kardiolodzy Spzoo, Włocławek
  - KO-MED Centra Kliniczne Spzoo KO-MED Centra Kliniczne Zamosc, Zamość
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Lecznej, Łęczna
- Portugal (9):
  - Hospital Garcia de Orta, EPE, Almada
  - Centro Hospitalar do Baixo Vouga, EPE - Hospital Infante Dom Pedro, Aveiro
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar e Universitario de Coimbra EPE, Coimbra
  - Hospital de Faro, EPE, Faro
  - Hospital da Senhora da Oliveira, Guimaraes, EPE, Guimarães
  - Associacao Protectora dos Diabeticos de Portugal, Lisbon
  - Unidade Local de Saude de Matosinhos - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital Casa de Saude Sao Mateus, Viseu
- Romania (11):
  - SC Centrul Medical de Diagnostic si Tratament Ambulator Neomed S.R.L, Brasov
  - Spitalul Clinic Universitar de Urgenta Elias, Bucharest
  - Institutul de Urgenţă pentru Boli Cardiovasculare "Prof. Dr. C. C. Iliescu",, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Cardiomed SRL, Craiova
  - Consultmed SRL, Iași
  - SC Cardiomed SRL, Iași
  - SC Endodigest SRL, Oradea
  - SC Sal Med SRL, Piteşti
  - Mediab SRL, Târgu Mureş
  - CMI Dr Podoleanu Cristian, Târgu Mureş
- Russia (41):
  - First City Clinical Hospital na E E Volosevich, Arkhangelsk
  - NSHI Departmental Hospital at the station Barnaul of OJSC Russian Railways, Barnaul
  - Regional State Budget Health care Institution Altay Regional Cardiology Dispensary, Barnaul
  - Regional Budget Healthcare Institution Cardiology Dispensary, Ivanovo
  - BHI of Republic Udmurtiya City clinical hospital 9 of Ministry of healthcare of Republic Udmurtiya, Izhevsk
  - FSBI Heart and Vessels Diseases complex problems Scientific Research Institution, Kemerovo
  - Kirov Regional State Budget Healthcare Institution Kirov City Clinical Hospital 1, Kirov
  - Regional Clinical Hospital 2 of the Ministry of Health Krasnodar region, Krasnodar
  - SBHI Scientific Research Institute Regional Clinical Hospital 1 named after S V Ochapovsky, Krasnodar
  - National Medical Research Center for therapy and preventive medicine, Moscow
  - Moscow SBHI City Clinical Hospital 15 n a O M Filatov of Moscow Healthcare Department, Moscow
  - SBHI of Moscow City clinical hospital 64 of Moscow Healthcare department, Moscow
  - City Clinical Hospital named after Zhadkevich, Moscow
  - FSBI Russian Cardiology Research and Production Complex, Moscow
  - SBHI of Nizhny Novgorod region Nizhny Novgorod regional clinical hospital na N A Semashko, Nizhny Novgorod
  - LLC RC Medical, Novosibirsk
  - SBHI of Novosibirsk Region City clinical hospital 1, Novosibirsk
  - FSBSI Scientific Research Institute of Therapy and preventive medicine, Novosibirsk
  - Budget Healthcare Institution of Omsk region Medical-sanitary unit 9, Omsk
  - Perm Regional Hospital for War Veterans, Perm
  - State Budget Institution of Ryazan Region Regional Clinical Hospital, Ryazan
  - City Polyclinic 27, Saint Petersburg
  - Saint Petersburg State Budget Healthcare Institution City Polyclinic 109, Saint Petersburg
  - City polyclinic 25 Nevsky district, Saint Petersburg
  - SBHI Medical and sports dispensary of Krasnogvardeisky district of Saint Petersburg, Saint Petersburg
  - Saint Petersburg SBHI City Hospital 38 named after N A Semashko, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Saint Petersburg State Budget Healthcare Institution Pokrovskaya City Hospital, Saint Petersburg
  - LLC Mart, Saint Petersburg
  - LLC Medinef Clinic, Sait-Petersburg
  - Samara Regional Clinical Cardiology Dispensary, Samara
  - Clinical Hospital named after S R Mirotvortsev, Saratov
  - Regional State Budget Helthcare Institution Smolensk Regional Clinical Hospital, Smolensk
  - State Budgetary Health Institution City Hospital 4 of the City of Sochi, Sochi
  - FSBSI Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk
  - Tyumen State Medical University, Tyumen
  - State Autonomous Healthcare Institution of the Tyumen region Medical Scientific Practical Center, Tyumen
  - SBHI of Vladimirskaya region City Hospital 4 of Vladimir, Vladimir
  - Family Medicine Clinic, Volgograd
  - Central City Clinical Hospital 1 of the Oktyabrsky District, Yekaterinburg
  - State Budget Medical Institution Sverdlovsk Regional Clinical Hospital N1, Yekaterinburg
- Slovakia (19):
  - Alian, sro, Bardejov
  - MediTask, sro, Bratislava
  - Narodny ustav srdcovych a cievnych chorob, as, Bratislava
  - Veria, sro, Bratislava
  - Nemocnica s poliklinikou Brezno, no, Brezno
  - Medical group Kosice sro, Košice
  - Cardio D and R, sro Kosice, Košice
  - Kardio 1 sro, Lučenec
  - Medi M and M sro, Moldava nad Bodvou
  - Oralek, sro, Námestovo
  - Kardiocentrum Nitra sro, Nitra
  - Kardiomed NZ, sro, Nové Zámky
  - Medikard, sro, Prešov
  - Medispol, sro, Prešov
  - Diab sro, Rožňava
  - Mediluk sro, Snina
  - Interna SK, sro, Svidník
  - Areteus sro, Trebišov
  - CardiOr, sro, Trenčín
- South Korea (19):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do
  - Yeungnam University Medical Center, Daegu
  - Keimyung University, Dongsan Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Ajou University Hospital, Suwon-si, Gyeonggi-do
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon-do
- Spain (25):
  - Hospital Virgen del Mar, Almería, Andalusia
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canarias, Canary Islands
  - Hospital Clinico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Equip Atencio Primaria Sardenya, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitari Sant Joan de Reus, Reus, Catalonia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Alvaro Cunqueiro, Vigo, Galicia
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario de La Princesa, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Infanta Sofia, Madrid
- Sweden (15):
  - Sodra Alvsborgs sjukhus, Borås
  - Falu Lasarett, Falun
  - Carlanderska, Gothenburg
  - Sahlgrenska Universitetssjukhus, Gothenburg
  - Obackakliniken i Harnosand, Härnösand
  - PharmaSite Helsingborg, Helsingborg
  - Lanssjukhuset Ryhov, Jönköping
  - Centralsjukhuset Karlstad, Karlstad
  - Skaraborgs sjukhus Lidkoping, Lidköping
  - Clemenstorgets Hjartmottagning, Lund
  - PharmaSite Malmo, Malmo
  - Ostersunds sjukhus, Östersund
  - Akardo MedSite, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Hallands sjukhus Varberg, Varberg
- Taiwan (10):
  - Hualien Tzu Chi Hospital, Hualien City, Hualien
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Mackay Memorial Hospital Tamsui Branch, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Ukraine (16):
  - Ivano-Frankivsk Regional Clinical Cardiology Center of Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Communal Healthcare Institution Kharkiv City Clinical Hospital No27, Kharkiv
  - Medical and Sanitary Unit of Open Joint Stock Company Kharkiv Tractor Plant, Kharkiv
  - Communal Noncommercial enterprise "City Hospital #8" of Kharkiv City Council, Kharkiv
  - Oleksandrivska Clinical Hospital of Kyiv, Kyiv
  - Kyiv City Clinical Hospital 1, Kyiv
  - Communal Noncommercial Institution Consultative and Diagnostic Center of Desnianskyi District of Kyi, Kyiv
  - Kyiv City Clinical Emergency Medical Care Hospital, Kyiv
  - National Scientific Center "M.D. Strazhesko Institute of Cardiology", Kyiv
  - State Institution National Scientific Center Acad MD Strazhesko Institute of cardiology of NAMS Ukr, Kyiv
  - State Institution National Scientific Center Acad Strazhesko Institute of Cardiology, Kyiv
  - Medical Centre CONSILIUM Medical, Kyiv
  - Zakarpattia Oblast Clinical Center of Cardiology and Cardio Surgery, Uzhhorod
  - Private Small Enterprise, Medical Center Pulse, Vinnytsia
  - Vinnytsia M I Pyrogov Regional Clinical Hospital Vinnytsia M I Pyrogov National Medical University, Vinnytsia
  - Communal Non-commercial enterprise "City Hospital #6 "of Zaporizhzhia City Council, Zaporizhzhia
- United Kingdom (50):
  - Aberdeen Royal Infirmary, Aberdeen
  - Barnsley Hospital, Barnsley
  - Royal United Hospital, Bath
  - Royal Victoria Hospital, Belfast
  - Ulster Hospital, Belfast
  - Ormeau Health Centre, Belfast
  - Bollington Medical Centre, Bollington
  - Royal Bournemouth Hospital, Bournemouth
  - West Walk Surgery, Bristol
  - University Hospitals of Derby and Burton NHS Foundation Trust, Burton-on-Trent
  - Ashgate Medical Practice, Chesterfield
  - Cleveleys Group Practice, Cleveleys
  - Lakeside Healthcare, Corby
  - Medinova Northamptonshire Dedicated Research Site, Corby
  - MeDiNova Warwickshire Quality Research Site, Coventry
  - Pound Hill Medical Group, Crawley
  - Ninewells Hospital, Dundee
  - Glasgow Royal Infirmary, Glasgow
  - Hull Royal Infirmary, Hull
  - Highlands Clinical Research Facility, Raigmore Hospital, Inverness
  - Royal Liverpool University Hospital, Liverpool
  - Barts Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Guys Hospital, London
  - Wythenshawe Hospital, Manchester
  - Medinova North London Dedicated Research Centre, Northwood
  - Nottingham City Hospital, Nottingham
  - George Eliot Hospital, Nuneaton
  - Medinova South London Dedicated Research Centre, Orpington
  - Mounts Bay Medical Hub, Penzance
  - The Health Centre Yaxley, Peterborough
  - The Adam Practice, Poole
  - Medinova East London Dedicated Research Centre, Romford
  - Sherbourne Medical Centre, Royal Leamington Spa
  - Eaton Socon Health Centre, Saint Neots
  - Ashfield Primary Care Centre, Sandbach
  - Scunthorpe General Hospital, Scunthorpe
  - Medinova Limited, Shipley
  - Lakeside Healthcare Stamford, Stamford
  - Lister Hospital, Stevenage
  - Singleton Hospital, Swansea
  - The Breckland Alliance, Thetford
  - Torbay Hospital, Torquay
  - Pinderfields Hospital, Wakefield
  - Sheepcot Medical Practice, Watford
  - Sandwell General Hospital, West Bromwich
  - Whitby Group Practice, Whitby
  - MeDiNova West London Quality Research Site, Wokingham
  - Worcestershire Royal Hospital, Worcester
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) The product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Bohula EA, Marston NA, Ruzza A, Murphy SA, De Ferrari GM, Diaz R, Leiter LA, Elliott-Davey M, Wang H, Bhatia AK, Giugliano RP, Sabatine MS. Rationale and design of the effect of evolocumab in patients at high cardiovascular risk without prior myocardial infarction or stroke (VESALIUS-CV) trial. Am Heart J. 2024 Mar;269:179-190. doi: 10.1016/j.ahj.2023.12.004. Epub 2023 Dec 29. PMID 38160917
- [Derived] Bohula EA, Marston NA, Bhatia AK, De Ferrari GM, Leiter LA, Nicolau JC, Park JG, Kuder JF, Murphy SA, Walsh E, Wang H, Blaha V, Budaj A, Cornel JH, Goudev A, Kiss RG, Lorenzatti AJ, Parkhomenko A, Cyrille M, Paiva da Silva Lima G, Ohman EM, Giugliano RP, Sabatine MS; VESALIUS-CV Investigators. Evolocumab in Patients without a Previous Myocardial Infarction or Stroke. N Engl J Med. 2026 Jan 8;394(2):117-127. doi: 10.1056/NEJMoa2514428. Epub 2025 Nov 8. PMID 41211925
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com